CLINICAL TRIAL: NCT00636103
Title: A Randomized Double-Blind Placebo-Controlled Study of the Effect of Traditional Chinese Medicines in the Treatment of Childhood Asthma
Brief Title: Efficacy Study of Herbal Formula CUF2 to Treat Childhood Asthma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University Grants Committee, Hong Kong (Other Government); Tuen Mun Hospital (Other Government)
Responsible Party: Rita Yn Tz Sung / Professor, Department of Paediatrics, The Chinese University of Hong Kong, Prince of Wales Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICM/CTS/002; AoE-10/01
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Asthma
Keywords: Traditional Chinese Medicine; Asthma; Paediatric
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CUF2 (Experimental)
  Interventions: Drug: CUF2
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CUF2 — 0.619g of dried aqueous extract of equal weights of 5 herbs (Astragalus mongholius Bunge, Cordyceps sinensis Sacc., Radix Stemonae, Bulbus Fritillariae Cirrhosae, Radix scutellariae).
  The dosage for children above 12 years old was three capsules twice daily and for children under 12 years old two capsules twice daily.
  Duration: 6 months
  Arms: CUF2
Other: Placebo — Dark coloured corn starch
  The dosage for children above 12 years old was three capsules twice daily and for children under 12 years old two capsules twice daily.
  Duration: 6 months
  Arms: Placebo

SUMMARY:
Asthma is a long-term disease process with genetic, allergic, environmental, infectious, emotional and dietary influences. The symptoms control are mainly using an inhaled drug, avoiding triggers or taking preventive medicine. Although side effects are unlikely at low dose of the asthma treatment, they have become apparent at the higher dose. Due to safety concern, parents often turn to complementary and alternative medicine which they believe is natural and safe and may help to reduce the conventional medication dosage.

There are number of reports that treatment with traditional Chinese herbs or formulas resulted in significant improvement in lung function and reduction in the airway hyper-reactivity reaction. Our study drug CUF2, was based on a classical formulae and had been proven to have anti-inflammatory and immunomodulatory activities in laboratory and animal studies.

With the pre-clinical evidence, this study aims to determine the effect of CUF2 on improving the clinical symptoms, biochemical markers, and requirement of steroid dosage among children with asthma.

DETAILED DESCRIPTION:
Patients are recruited from 2 major governmental hospitals in Hong Kong (Prince of Wales Hospital and Tuen Mun Hospital),aged between 7 to 15 years with mild to moderate asthma according to the Global Initiative for Asthma guideline, on regular inhaled steroid therapy and capable to perform a lung function test.

However, those patients are excluded if they could not swallow capsules or had received parenteral or oral corticosteroids, nedocromil, cromolyn, theophylline or anticonvulsants in the past 4 weeks.

Before study start, written informed consent will be obtained from each patient and one of their parents. The eligible patients will be randomly assigned to receive CUF2 or placebo capsules for 6 months. For the dosage, children aged above 12 years old, 3 capsules twice daily and under 12 years old, 2 capsules twice daily.

During the 6 months period, below measurements will be taken:

* The severity of asthma symptoms was assessed using a modified Disease Severity Score (DSS)
* Lung Function Test by spirometry (SpiroPro Jaeger Toennies, Hoechberg, Germany)
* Conventional Medication consumption, according to GINA/NIH guidelines.
* Blood test, EDTA and clotted blood samples were taken at the baseline and end of the study for eosinophil counts, IgE level and cytokine assay.

ELIGIBILITY:
Inclusion Criteria:

* Persistent Mild to Moderate Asthma
* Aged 7 to 15 years
* On Regular inhaled steroid therapy
* Able to perform reproducible spirometry

Exclusion Criteria:

* Could not swallow capsules
* Received parenteral or oral corticosteroids, nedocromil, cromolyn, theophylline or anticonvulsants in past 4 weeks

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2002-07; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Reduction of steroid dosage | 6 months

SECONDARY OUTCOMES:
Asthma symptoms | 6 months
Lung function test | 6 months
Biochemical markers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rita YT Sung, MD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of Paediatrics, Prince of Wales Hospital, Hong Kong
  - Department of Paediatrics, Tuen Mun Hospital, Hong Kong

REFERENCES:
- [Background] Leung R, Wong G, Lau J, Ho A, Chan JK, Choy D, Douglass C, Lai CK. Prevalence of asthma and allergy in Hong Kong schoolchildren: an ISAAC study. Eur Respir J. 1997 Feb;10(2):354-60. doi: 10.1183/09031936.97.10020354. PMID 9042632
- [Background] Lau YL, Karlberg J. Prevalence and risk factors of childhood asthma, rhinitis and eczema in Hong Kong. J Paediatr Child Health. 1998 Feb;34(1):47-52. doi: 10.1046/j.1440-1754.1998.00217.x. PMID 9568941
- [Background] Rao R, Gregson RK, Jones AC, Miles EA, Campbell MJ, Warner JO. Systemic effects of inhaled corticosteroids on growth and bone turnover in childhood asthma: a comparison of fluticasone with beclomethasone. Eur Respir J. 1999 Jan;13(1):87-94. doi: 10.1183/09031936.99.13108799. PMID 10836329
- [Background] But P, Chang C. Chinese herbal medicine in the treatment of asthma and allergies. Clin Rev Allergy Immunol. 1996 Fall;14(3):253-69. doi: 10.1007/BF02802218. No abstract available. PMID 8932956
- [Background] Hsieh KH. Evaluation of efficacy of traditional Chinese medicines in the treatment of childhood bronchial asthma: clinical trial, immunological tests and animal study. Taiwan Asthma Study Group. Pediatr Allergy Immunol. 1996 Aug;7(3):130-40. doi: 10.1111/j.1399-3038.1996.tb00120.x. PMID 9116877
- [Background] Critchley JA, Zhang Y, Suthisisang CC, Chan TY, Tomlinson B. Alternative therapies and medical science: designing clinical trials of alternative/complementary medicines--is evidence-based traditional Chinese medicine attainable? J Clin Pharmacol. 2000 May;40(5):462-7. doi: 10.1177/00912700022009224. PMID 10806598
- [Background] Lin LZ, He XG, Lindenmaier M, Nolan G, Yang J, Cleary M, Qiu SX, Cordell GA. Liquid chromatography-electrospray ionization mass spectrometry study of the flavonoids of the roots of Astragalus mongholicus and A. membranaceus. J Chromatogr A. 2000 Apr 21;876(1-2):87-95. doi: 10.1016/s0021-9673(00)00149-7. PMID 10823504
- [Background] Patocka J. Anti-inflammatory triterpenoids from mysterious mushroom Ganoderma lucidum and their potential possibility in modern medicine. Acta Medica (Hradec Kralove). 1999;42(4):123-5. PMID 10812678
- [Background] Cheong J, Jung W, Park W. Characterization of an alkali-extracted peptidoglycan from Korean Ganoderma lucidum. Arch Pharm Res. 1999 Oct;22(5):515-9. doi: 10.1007/BF02979162. PMID 10549581
- [Background] Kong XT, Fang HT, Jiang GQ, Zhai SZ, O'Connell DL, Brewster DR. Treatment of acute bronchiolitis with Chinese herbs. Arch Dis Child. 1993 Apr;68(4):468-71. doi: 10.1136/adc.68.4.468. PMID 8503668
- [Background] Standards for the diagnosis and care of patients with chronic obstructive pulmonary disease (COPD) and asthma. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, November 1986. Am Rev Respir Dis. 1987 Jul;136(1):225-44. doi: 10.1164/ajrccm/136.1.225. PMID 3605835
- [Derived] Wong EL, Sung RY, Leung TF, Wong YO, Li AM, Cheung KL, Wong CK, Fok TF, Leung PC. Randomized, double-blind, placebo-controlled trial of herbal therapy for children with asthma. J Altern Complement Med. 2009 Oct;15(10):1091-7. doi: 10.1089/acm.2008.0626. PMID 19821718